CLINICAL TRIAL: NCT05629156
Title: Injury and Illness Surveillance At the FIFA World Cup Qatar 2022TM
Acronym: IISFWC22
Status: Completed | Type: Observational
Sponsor: Federation Internationale de Football Association (Other)
Collaborators: Aspetar Orthopaedic and Sports Medicine Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Injuries; Illness Physical; Illness, Mental
MeSH Terms: conditions — Wounds and Injuries; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention implemented. Observational study only — Observational study only. Injuries and illnesses and exposure is registered using standardized paper forms.

SUMMARY:
The project aims to provide an overview of injury and illnesses during the FIFA World Cup Qatar 2022. All teams are invited to participate and record details on time-loss injury and illness occurrence and training and match exposure during the tournament. In order to assess the severity of injuries (based on the length of time a player is unable to play for), all injuries are to be monitored until they are fully rehabilitated, even if this is after the end of the tournament. This information will be recorded by the team physicians and provided on daily report forms to the research team. Data will be encrypted before analysis and only anonymized data will be published. Descriptive statistics are used to provide an overview of the participant demographics and injury and illness occurrence. Injury incidence is calculated as number of injuries per 1000 hours of exposure, and injury burden is calculated as time-loss days per 1000 hours of exposure. Injury incidence and burden will be reported for training and match injuries separately. Illness incidence is calculated per 365 exposure days.

DETAILED DESCRIPTION:
Background Injury rates in football are closely associated with team performance. Teams are more likely to lose matches in which they have suffered injuries, and teams with fewer injuries have significantly better results both in international tournaments and in national leagues. Injuries can have both high short- and long-term consequences for an individual player's health and career. Illness rates in professional football is lower than injury rates, but it is unclear whether illness rates are higher in international tournaments, which often include travel, exposure to different environments, high match significance, and match congestion.

Injury surveillance is a cornerstone in the development of injury prevention programs. Injury and illness prevention strategies are continuously being developed and improved, and it is therefore important with ongoing surveillance. Additionally, there has been scientific advances in methodology, which can ensure more detailed and accurate information.

Objectives The primary objective is to provide an overview of the incidence and characteristics of time-loss injuries and illnesses during the FIFA World Cup Qatar 2022.

The primary variables of interest are time-loss injuries and time-loss illnesses.

* Time-loss is defined as inability of a player to complete the current or future training session or match.
* Injury is defined as tissue damage or other derangement of normal physical function resulting from rapid or repetitive transfer of kinetic energy.
* Illness is defined as a health-related complaint or disorder experienced by an athlete, not considered as an injury.

A secondary aim is to analyse injury mechanisms through match video footage of the observed time-loss injuries.

Design Prospective observational cohort study.

This research project will be performed at the FIFA World Cup Qatar 2022, which is played November 20th and December 18th, 2022 in Qatar.

Study duration The study will start from the first day of training with the national team prior the tournament until the day of the last match of the tournament. Consequently, the number of recordings will vary between teams depending on the duration of their pre-tournament training (usually 1-3 weeks), and their performance and progression through the tournament. In order to assess the severity of injuries (based on the length of time a player is unable to play for), all injuries are to be recorded until they are fully rehabilitated, even if this is after the end of the tournament. Each contact person therefore also needs to report when an injured player who has left the tournament has returned to full training with their club team after the tournament.

Demographic information Individual demographic information, including age, height, weight, playing position, and leg dominance (preferred kicking leg), is collected following inclusion.

Injury & illness registration Data on injury and illness is gathered following the recommended methodology in the football extension of the International Olympic Committee consensus statement on methods for recording and reporting of epidemiological data on injury and illness in sport. This includes characteristics such as mode of onset, injury mechanism, diagnosis and classification according to body area, tissue, and pathology type, and illness categories for organ system and etiology. Time-loss will be counted in number of days.

Exposure registration Training and match exposure will be recorded in minutes for each participant for the duration of the tournament. Training exposure includes for example any sports-specific training, strength and conditioning sessions, and active recovery sessions. Illness exposure will be recorded in days for each participant from their first day of training until their last match.

Descriptive statistics is used to provide an overview of the participant demographics and injury and illness occurrence. Injury incidence is calculated as number of injuries per 1000 hours of exposure, and injury burden is calculated as time-loss days per 1000 hours of exposure. Injury incidence and burden will be reported for training and match injuries separately. Illness incidence is calculated per 365 exposure days. Potential missing data will be excluded from analysis and reported accordingly.

Sample size No a priori sample size calculation is performed as we will attempt to include all eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* All participating football players at the FIFA World Cup Qatar 2022.

Exclusion Criteria:

* No exclusion criteria are present except declining to provide consent for data to be used in this study.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The FIFA World Cup Qatar 2022 includes 32 national teams, and each team is allowed to select 26 players, giving at total of 832 potential participants. In total, 64 matches will be played over 29 days.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence and burden of Time-loss injuries | November-December 2022
  Time-loss is defined as inability of a player to complete the current or future training session or match.
  Injury is defined as tissue damage or other derangement of normal physical function resulting from rapid or repetitive transfer of kinetic energy.
Incidence and burden of Time-loss illnesses | November-December 2022
  Time-loss is defined as inability of a player to complete the current or future training session or match.
  Illness is defined as a health-related complaint or disorder experienced by an athlete, not considered as an injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Aspetar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No